CLINICAL TRIAL: NCT07248462
Title: Integrating Mental Health and Neglected Tropical Disease Interventions to Support Equitable People-Centred Care in Ghana
Brief Title: Integrating Mental Health Into Neglected Tropical Disease Care in Ghana
Acronym: IMAGINE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Liverpool School of Tropical Medicine (Other)
Collaborators: University of Health and Allied Sciences, Ho (Unknown); Fundación Anesvad (Unknown); Effect:Hope (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 25-026
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Leprosy; Lymphatic Filariases; Buruli Ulcer; Onchocerciasis; Yaws
MeSH Terms: conditions — Leprosy; Elephantiasis, Filarial; Buruli Ulcer; Onchocerciasis; Yaws | interventions — Mental Health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Persons affected by NTDs (Experimental): Persons affected by NTDs in 4 areas in Ghana (Ho, Hohoe, Bole and Ellembele)
  Interventions: Other: WHO Essential Care package for mental health and NTDs

INTERVENTIONS:
Other: WHO Essential Care package for mental health and NTDs — Participants will receive integrated mental health and NTD care, following the WHO essential care package, using a stepped-care model with interventions at different levels of the health system. There will be population and community-level initiatives (e.g. peer support groups, awareness raising), decentralised management of patients including health worker capcity strenghtening (e.g. mhGAP, screening as part of routine care), and referral into secondary or tertiary care.

SUMMARY:
Background Neglected Tropical Diseases (NTDs) are a group of diseases that are more common among the poorest people in the poorest countries. People affected by these conditions often experience pain, changes in their physical appearance, stigma and discrimination. As a result, they are more likely to experience mental distress including depression and anxiety. It is important that people affected by these conditions are found early, so that they can start treatment to stop the progression of the condition and to support their mental wellbeing. The World Health Organisation recently developed guidance that explains more about including mental health awareness and care as part of the management of people who have these conditions. This is called the Essential Care Package for NTDs, Stigma and Mental Health Conditions. However, so far there has been limited research about 'what works' when providing this package to people who need it.

Aim of the study Through this study, we aim to understand 'How can the health system in Ghana provide the essential care package for people affected by skin NTDs for large groups of the population (at scale)?; and how to do this in a way that means everyone can access it (that is fair) and that is effective (works well)?'

Methods/ Design In order to do this, we will develop a Ghanaian version of the Essential Care Package and associated resources to support its implementation. We will do this by including people affected by NTDs to help us understand the needs and priorities from their perspective. Working together with researchers, health workers and those who make decisions about health, people affected will be supported to identify their priorities and to take part in developing what will be included in this Ghanaian ECP. This will happen by using creative forms of research that encourage people to participate and through the process, with workshops to include their opinions scheduled throughout.

Once this has been developed the Government will then start to introduce the Ghanaian ECP in selected study districts. At the same time, we will monitor and evaluate what is happening to understand what parts work well? who they work best for? in what settings? and for how long? We will carry out different types of research to understand who has access to this new package of services? (how fair is it?), how well it works? How the health workers and health system take up and use the new ECP? How the new ECP is rolled out and introduced as part of the health system? And whether it can be maintained and continue beyond the end of the study?

Discussion Through this study, we hope that people affected by NTDs and mental health conditions will be able to access and use quality health services when they need them; that communities will have a better understanding about NTDs and mental health conditions; and that government departments will work better together to provide care for NTDs and mental health conditions together.

ELIGIBILITY:
Inclusion Criteria:

* Affected by one of the target NTDs (leprosy, LF, buruli Ulcer, Yaws, Onchocersiasis)
* Living in one of the intervention areas (Bole, Ho, Hohoe, Ellembele)
* Aged 18 years and above

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Depression | From enrolment to the end of the intervention period 12 months later
  Depression as measured by PHQ-9
anxiety | From enrolment until end of intervention period 12 months later
  Anxiety as measured by GAD-7
Mental wellbeing | From enrolment until end of intervention period 12 months later
  Mental wellbeing as measured by Warwick mental wellbeing scale

SECONDARY OUTCOMES:
Quality of Life | From enrolment until end of intervention period 12 months later
  QoL as measured by EQ-5D-5L
Participation | From enrolment until end of intervention 12 months later
  Social participation as measured by Participation Scale
Stigma | Enrolment - end of intervention period 12 months later
  Stigma as measured by sari stigma scale

REFERENCES:
- See also: Related Info — https://uhas.edu.gh/uhas/blog/uhas-ntds-centre-uses-imagine-ghana-project-target-mental-health-and-tropical-disease-care

DOCUMENTS (1):
  • Study Protocol (2025-10-30): https://cdn.clinicaltrials.gov/large-docs/62/NCT07248462/Prot_000.pdf